CLINICAL TRIAL: NCT05711043
Title: The GATE Trial: Endoscopic Sutured Gastroplasty in Type 2 Diabetic, Obese Patients Using the Endomina Device - a Randomized Controlled Trial
Brief Title: The GATE Trial: Endoscopic Sutured Gastroplasty in Type 2 Diabetic, Obese Patients Using the Endomina Device
Acronym: GATE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Fenna Beeren, Coordinating researcher, Radboud University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL83606.091.23
Record Dates: First submitted 2023-01-23; First posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-02

CONDITIONS: Diabetes Mellitus Type 2 in Obese

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Endoscopic sutured gastroplasty with endomina device
  Interventions: Device: Endoscopic sutured gastroplasty with endomina
- Control group (No Intervention): Standard diabetes care

INTERVENTIONS:
Device: Endoscopic sutured gastroplasty with endomina — Subjects in the intervention group will be treated with an ESG with the endomina ® and TAPES devices (Endo Tools Therapeutics S.A.), both CE-marked for endoscopic gastroplasty. The endomina is a device that can be attached to an endoscope and allows remote actuation of the device during a peroral intervention. Thanks to a therapeutic channel that can be angled perpendicularly to the axis of vision of the endoscope, it allows the possibilities of making transoral full thickness tissue apposition and performing, via a transoral route, large plications with tight serosa to serosa apposition in the stomach. This suturing will be done from the incisura to the upper body of the stomach, along the great curvature with TAPES, a single use needle preloaded with suture.
  In addition to the endomina device, any other required endoscopic accessories can be used during the procedure (e.g., grasping forceps, loop cutter).
  Other Names: ESG; Endoscopic sleeve gastrectomy; Endomina
  Arms: Intervention group

SUMMARY:
Rationale: Diabetes mellitus is a chronic disease that is often associated with long-term macrovascular and microvascular complications and decreased life expectancy. Approximately 70% of patients with type 2 diabetes mellitus (DM2) are overweight or obese. Weight loss benefits several aspects of DM2, such as improved glycemic control, increased insulin sensitivity and reduced fasting insulin. Interventions for weight loss in patients with DM2 include diet, exercise, but also pharmacotherapy and bariatric surgery.

Bariatric surgery is indicated at a body mass index (BMI) > 35 kg/m², in combination with other comorbidities. It is associated with better glycemic control and more weight reduction, compared to intensive medical treatment alone. For patients with not adequately controlled DM2 who are not eligible for surgery (i.e., BMI of < 35 kg/m²), there is a therapeutic gap, which could be filled by one of the currently available endoscopic therapies aiming to reduce weight. One of these therapies is endoscopic sutured gastroplasty (ESG), performed with the endomina device (EndoTools Therapeutics S.A.). There is however a paucity of data showing the effect of ESG on metabolic comorbidities including DM2. We hypothesize that ESG with the endomina device will improve glycemic control in patients with DM2 and obesity.

Objective: To evaluate the efficacy of ESG with the endomina device on glycemic control, in obese insulin treated type 2 diabetic patients.

Study design: This is a prospective, randomized controlled trial. Study population: 58 subjects (29 in each group) with a BMI between 30 and 40 kg/m² and DM2, treated with insulin therapy.

Intervention (if applicable): The intervention group will receive ESG performed with the endomina device. The control group will receive standard diabetic care.

Main study parameters/endpoints: The primary endpoint is the proportion of patients with a clinically relevant reduction of insulin dose. Secondary endpoints include among others reduction in HbA1c, remission of diabetes, weight loss, quality of life and (serious) adverse events.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: An ESG with the endomina device is known to have only minor adverse events (transient abdominal cramps, nausea, vomiting), and a serious adverse event rate of <1% (no surgical intervention needed, no mortality).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-65 years
* Diagnosed with DM2

  * since at least 1 year
  * currently under stable dose of insulin for at least 6 months
  * with or without use of any other oral glucose lowering medication (e.g., metformin, glucagon-like peptide (GLP)-1 receptor agonist)
* HbA1c level of 7.0-11.0% (53-75 mmol/mol) prior to inclusion
* BMI of 30-40 kg/m²
* Must be able to comply with all study requirements for the duration of the study as outlined in the protocol (including compliance to treatment, dietary follow up, visits as scheduled and all study specific procedures)
* Must be able to understand and be willing to provide written informed consent
* Must be eligible for general anesthesia or deep sedation with propofol

Exclusion Criteria:

* Achalasia and any other esophageal motility disorders
* Severe esophagitis (grade C or D)
* Gastro-duodenal ulcer
* Gastrointestinal stenosis or obstruction
* Any history of esophageal or gastric surgery
* Heart diseases: unstable angina, myocardial infarction within the past year, or heart disease classified within the New York Heart Association's Class III or IV functional capacity
* Uncontrolled hypertension (systolic blood pressure >180 mm Hg and/or diastolic blood pressure >100 mm Hg under medication) during last 3 months;
* Severe renal, hepatic, pulmonary disease or cancer (cancer in the past 5 years, except basal cell carcinoma)
* Known with, or history of, eating disorder
* Pregnancy, breast feeding or desire to become pregnant in the coming 12 months
* Any previous bariatric surgery, or endoscopic obesity-related intervention (including Primary Obesity Surgery Endoscopic (POSE), OverStitch, etc.). Intragastric balloon removed within the last 6 months
* Planned gastric surgery 60 days post intervention
* Anticoagulant therapy that cannot be temporarily stopped at the time of the procedure.
* Currently participating in another study (involving change of treatment).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with a clinically relevant reduction of insulin dose after 12 months | 12 months
  A clinically relevant reduction is defined as a 50% dose reduction.

SECONDARY OUTCOMES:
Rate of Serious Adverse Events (SAE) and Serious Adverse Device Effects (SADE) during and post procedure at 12 months | 1 year
(Serious) adverse events up to 1-month follow-up for subjects undergoing the procedure under procedural sedation with propofol | 1 month
Cardiovascular events (stroke/Transient Ischemic Attack (TIA), myocardial infarction, admission for heart failure) after 12 months | 1 year
All-cause mortality after 12 months | 1 year
Reduction in HbA1c after 1 month, 3-, 6-, and 12-months follow-up | 1 year
Proportion of subjects with a clinically relevant reduction of insulin dose after 1 month, 3 and 6 months. | 6 months
Proportion of subjects with a clinically relevant decrease in HbA1c after 1 month, 3-, 6-, and 12-months follow-up. A clinically relevant decrease in HbA1c is defined as 2.6% (5mmol/mol). | 1 year
Reduction in fasting plasma glucose levels after 1 month, 3-, 6-, and 12-months follow-up. | 1 year
Proportion of subjects with reduced number and/or reduced dose(s) of (oral) glucose lowering medication after 1 month, 3-, 6-, and 12-months follow-up. | 1 year
Proportion of subjects with remission of diabetes after 6, 9 and 12 months. Remission is defined as HbA1c < 6.5% (48 mmol/mol), fasting glucose of < 5.6 mmol/l without glucose-lowering medication for at least 3 months. | 1 year
Proportion of subjects with mean % excess weight loss (%EWL) of more than 25% after 1 month, 3-, 6-, and 12-months follow-up. | 1 year
%EWL after 1 month, 3-, 6-, and 12-months follow-up. | 1 year
Proportion of subjects with mean % total body weight loss (%TBWL) of more than 5% after 1 month, 3-, 6-, and 12-months follow-up. | 1 year
%TBWL after 1 month, 3-, 6-, and 12-months follow-up. | 1 year
Decrease in blood pressure after 1 month, 3-, 6-, and 12-months follow-up. | 1 year
EuroQol 5Dimension 5Level (EQ-5D-5L) after 1 month, 3-, 6-, and 12-months follow-up. | 1 year
Diabetes Treatment Satisfaction Questionnaire (DTSQ) after 1 month, 3-, 6-, and 12-months follow-up. | 1 year
Costs | 1 year
  Costs include health care recourses used (including intervention, endomina device and TAPES, hospital admissions, visits to specialists and general practitioner, emergency room visits, medications used), costs for insulin therapy (including medication, administration, glycemia measurement material)
Cost-effectiveness | 1 year
  Using quality adjusted life years (QALYs)

CONTACTS AND LOCATIONS:
Locations (1):
- Rijnstate, Arnhem, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Upon request after publication
Supporting Information: Study Protocol, SAP, CSR